CLINICAL TRIAL: NCT00467662
Title: The Safety, Efficacy and Convenience of Use of the Natural Agent "Superlysin Gel" as Treatment for Herpes Labialis in Comparison to Acyclovir 5% and Docozanole 10%.
Brief Title: Comparison of Topical Antiviral Agents for Labial Cold Sores (Herpes Labialis)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 376.hmo-ctil
Record Dates: First submitted 2007-04-17; First posted 2007-05-01 (Estimated); Last update posted 2007-05-01 (Estimated); Status verified 2007-04

CONDITIONS: Reccurent Herpes Labialis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Acyclovir 5%
Drug: Docosanol 10%
Device: Superlysine gel

SUMMARY:
Recurrent cold sores - herpes simplex labialis (HSL) occurs in 20-40% of the US population and patient seek treatment because of the discomfort and visibility of the lesion although it is a self limiting disease. The purpose of this study is to check the safety, Efficacy and convenience of Use of the Natural Agent "Superlysin Gel" as Treatment for Herpes Labialis in Comparison to Acyclovir 5% and Docozanole 10%.

DETAILED DESCRIPTION:
Study design:

-Double blinded non-inferiority prospective parallel-group, intend to treat trial. Enrolment of 75 patients (25 randomized for each group). - Approval of the Institutional Ethical Review Board -

Study design:

- Patient characteristics (selected) and historical information assessment including: Race, average episode duration from patient history Duration of most recent previous episode Time since last onset of oral-facial herpes simplex Time since first onset of oral-facial herpes simplex Does patient experience localized prodrome?

* Experiment duration; 5 to 10 days
* 4 visits (days 1, 3,6,10)
* 5 application /day for each derivative
* Documentation Metric digital images of localized area signs at each visit Clinical assessment of prodrome/erythema, papule, vesicle, ulcer, crust, or healed skin (with or without residual erythema) Visual analogue scale (VAS) for subjective assessment of pain, burning, itching or tingling at each visit
* Calculation of primary efficacy end point (time to healing); from the date and time of the initiation of therapy until the date and time of the clinic visit at which complete resolution of all local signs and symptoms, i.e. the lesion had aborted or complete healing had occurred (censored at day 10)

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent
* Age range (yrs) 18-70
* Gender ; Males and females
* Health status; immuno-competent
* Clinical history of HSL with at least two recurrences during the past 12 months. The most recent previous episode must have healed at least 14 days before screening.
* Less than 12 hours after prodrome initiation (i.e. local erythema w/o blistering, tingling and or burning sensation, soreness)

Exclusion criteria:

* Pregnant women
* Mentally disabled
* No intra-oral lesions, or lesions above the nostrils and below the chin
* No topical steroid use and no systemic antiviral current treatments within 7 days before the study
* No known allergies to topical cosmetics
* No use cosmetics on or around the mouth during the treatment period
* No concomitant use of systemic corticosteroids or other drugs known to induce immune stimulation or immune suppression

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)

PRIMARY OUTCOMES:
Reducing healing process and duration of cold sores using superlysin gel

CONTACTS AND LOCATIONS:
Overall Officials: Doron Aframian, DMD,PhD, Study Chair — Salivary Gland Clinic, Department of Oral Medicine The Hebrew University-Hadassah School of Dental Medicine Jerusalem, Israel P.O.B 12272, Zip code 91120